CLINICAL TRIAL: NCT00513903
Title: Enhanced Continuity of Pharmacy Care for Cardiovascular or Pulmonary Diseases
Brief Title: Expanding the Role of Pharmacists in Treating Persons With Cardiovascular or Lung Diseases
Acronym: IowaCOC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 498; R01HL082711 (NIH); R01HL082711-01A2 (NIH)
Record Dates: First submitted 2007-08-07; First posted 2007-08-09 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Cardiovascular Diseases; Lung Diseases
Keywords: Pulmonary Diseases; Continuity of Pharmacy Care
MeSH Terms: conditions — Cardiovascular Diseases; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Minimal intervention (Active Comparator): Minimal intervention group patients will be seen by a clinical pharmacist in the hospital but will not receive followup after hospital discharge.
  Interventions: Behavioral: Minimal intervention
- Enhanced intervention (Experimental): Enhanced intervention patients will receive care from a clinical pharmacist during hospitalization and followup by phone after hospitalization.
  Interventions: Behavioral: Enhanced Intervention
- Control (No Intervention): Control arm patients will not be seen by the clinical pharmacist.

INTERVENTIONS:
Behavioral: Minimal intervention — Minimal intervention patients will be seen by a clinical pharmacist during the hospitalization period to improve continuity of pharmacy care following hospital discharge.
  Arms: Minimal intervention
Behavioral: Enhanced Intervention — Enhanced intervention patients will be visited in the hospital and will also be called by the clinical pharmacist following discharge to follow-up on any problems that might have developed after discharge.
  Arms: Enhanced intervention

SUMMARY:
This study will test whether enhanced continuity of pharmacy care that includes increased communication between inpatient and outpatient settings will improve the appropriateness of medication therapy and reduce the number of serious adverse drug events, hospitalizations and unscheduled office visits in vulnerable patients with cardiovascular disease, pulmonary disease or diabetes.

DETAILED DESCRIPTION:
Drugs used to treat cardiovascular and lung diseases are the most frequent cause of hospitalizations and emergency department visits related to inadequate therapy or ADEs. ADEs occur in 25% of patients who are able to walk and may cause up to 17% of hospital admissions among the elderly. A lack of communication and coordination between the hospital setting and the patient's own community setting, upon patient discharge, may contribute to the high number of ADEs. By expanding the role of pharmacists and encouraging communication between hospitals and pharmacists, the number of ADEs may be reduced. There have been a few small studies that have examined the way patient information is transferred between hospital and community pharmacists, but these studies did not involve the patients' primary care physicians nor did they fully evaluate the effect of communication between hospital and community pharmacists. The purpose of this study is to evaluate the effectiveness of providing a pharmacist case manager to hospitalized patients with cardiovascular or lung disease at reducing the number of ADEs, re-hospitalizations, and unscheduled medical visits.

This study will enroll individuals with certain conditions or diseases who are admitted to the hospital. Participants will be randomly assigned to either a control group, a minimal treatment group, or an enhanced treatment group. Participants in the minimal and enhanced treatment groups will meet with a pharmacist case manager while in the hospital to conduct a medication history review. The case manager will also meet with participants at the time of hospital discharge and provide them with a discharge summary and educational materials. Additionally, for participants in the enhanced treatment group, the case manager will do the following: transfer the discharge summary data to the participant's community physician and pharmacist; call the participant 3 to 5 days following discharge from the hospital and as needed thereafter to resolve medication problems; and communicate with and make recommendations to the participant's community physician and pharmacist. All participants will meet with a study research nurse immediately after study entry to complete questionnaires. Study nurses will also call all participants 30 and 90 days following hospital discharge to collect adverse event information. Surveys will be completed by each participant's pharmacist and primary care physician 90 days following the participant's discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Speaks either English or Spanish
* Willing to obtain all long-term prescriptions from one community pharmacy during the 90-day study period
* Diagnosed with at least one of the following conditions: high blood pressure, hyperlipidemia, heart failure, coronary artery disease, heart attack, stroke, transient ischemic attack, asthma, chronic obstructive pulmonary disease (COPD), diabetes, or receiving oral anticoagulation therapy
* Admitted to the general medicine, family medicine, cardiology, or orthopedics services hospital department

Exclusion Criteria:

* Does not have a working telephone
* Has a hearing impairment that does not allow the use of a telephone
* Enrolled in Iowa Care (i.e., individual has no community physician or community pharmacist following hospital discharge)
* Life expectancy estimated at less than 6 months at the time of study entry
* Dementia or cognitive impairment
* Severe psychiatric or psychosocial factors, including substance abuse, that may impair the desire or ability to complete all aspects of the study
* Admission to the psychiatric, surgery, or hematology/oncology services hospital department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 954 (Actual)
Dates: Start 2008-03; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
ADEs | Measured 30 and 90 days after hospital discharge
Medication appropriateness | Measured 30 and 90 days after hospital discharge by the Hanlon et al. Medication Appropriateness Index
Complications related to medications, including the number of hospital readmissions, unscheduled visits to emergency departments or urgent care facilities, and physician visits related to a medication problem or ADE | Measured 30 and 90 days after hospital discharge
Cost-effectiveness of the minimal or enhanced treatment compared to usual care | Measured 30 and 90 days after hospital discharge

SECONDARY OUTCOMES:
Number of medications | Measured 30 and 90 days after hospital discharge
Complete medication list | Measured 30 and 90 days after hospital discharge
Community physician and pharmacist surveys | Measured 90 days after participant's hospital discharge
Medication adherence | Measured 30 and 90 days after hospital discharge
Barriers to patient adherence | Measured at baseline by scores on the following questionnaires: self-efficacy, cognitive impairment (Pfeiffer Mental Status Questionnaire), medication management skills and the Katz index of activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Barry L. Carter, PharmD, Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Carter BL, Farris KB, Abramowitz PW, Weetman DB, Kaboli PJ, Dawson JD, James PA, Christensen AJ, Brooks JM. The Iowa Continuity of Care study: Background and methods. Am J Health Syst Pharm. 2008 Sep 1;65(17):1631-42. doi: 10.2146/ajhp070600. PMID 18714110
- [Result] Farley TM, Shelsky C, Powell S, Farris KB, Carter BL. Effect of clinical pharmacist intervention on medication discrepancies following hospital discharge. Int J Clin Pharm. 2014 Apr;36(2):430-7. doi: 10.1007/s11096-014-9917-x. Epub 2014 Feb 11. PMID 24515550
- [Result] Israel EN, Farley TM, Farris KB, Carter BL. Underutilization of cardiovascular medications: effect of a continuity-of-care program. Am J Health Syst Pharm. 2013 Sep 15;70(18):1592-600. doi: 10.2146/ajhp120786. PMID 23988600
- [Result] Anderegg SV, Demik DE, Carter BL, Dawson JD, Farris K, Shelsky C, Kaboli P. Acceptance of recommendations by inpatient pharmacy case managers: unintended consequences of hospitalist and specialist care. Pharmacotherapy. 2013 Jan;33(1):11-21. doi: 10.1002/phar.1164. PMID 23307540
- [Derived] Farris KB, Carter BL, Xu Y, Dawson JD, Shelsky C, Weetman DB, Kaboli PJ, James PA, Christensen AJ, Brooks JM. Effect of a care transition intervention by pharmacists: an RCT. BMC Health Serv Res. 2014 Sep 18;14:406. doi: 10.1186/1472-6963-14-406. PMID 25234932